Official title of the study: Life-Skills Training Program: Its effect on Selfefficacy among Patients with Substance Use Disorders

**NCT number: Pending** 

Date of the document: 1/4/2023

Substance use disorders is episodic, with periods of abstinence, reduction of use, and relapse as the prevailing pattern, often with the course of events being influenced by external factors such as the availability of drugs and societal

pressures (Sapkota, et al., 2019)

Self-Efficacy (SE) plays an essential role in the maintenance of abstinence

from drugs and alcohol which is a belief regarding one's ability to successfully

resist performing a behavior, and outcome expectancies, meaning the anticipated

consequences of performing a behavior (Alanazi, et al., 2022). Also, Abstinence

self-efficacy (ASE) as the belief individuals have in their ability to abstain from

engaging in an undesired action. ASE includes an individual's level of confidence

with their ability to abstain from substances for an extended period of time (Niles,

et al., 2022).

Overall, Self-efficacy addresses the individual's perception of control of

life events and is predictive of a person's goals and performance and affected with

negative things such as shame (Bahramabadian, Mojtabaie, & Sabet, 2021).

Life skills are defined as a group of psychosocial competencies and

interpersonal skills that help people make informed decisions, solve problems,

think critically and creatively, communicate effectively, build healthy

relationships, empathize with others, and cope with and manage their lives in a

healthy and productive manner (UNODC, 2023).

Life skills may be directed toward personal actions or actions toward

3

others, as well as toward actions to change the surrounding environment to make it

conducive to health (WHO, 2023). Bearing the WHO definition in mind, the Basic

Life Skills curriculum offers youth the emotional, social, and intellectual tools

needed to achieve success in life – on personal level, interpersonal level, also,

within their community and workplaces (UNICEF. 2023)

Drug users often have problems with social and interpersonal relationships.

The lack of adequate social relationships for patients' will should various

negative personal and social consequences for patients' health, their families,

friends, and society. Life skills training could effectively improve their social

communication with parents, family, and friends. Life skills training should be part

of addiction prevention training programs (Ebrahem, Radwan, & El Amrosy,

2022).

Life-skills training program designed to prevent substance use relapse which

typically combine training about self-management skills (e.g., coping with stress),

social skills (e.g., assertiveness), and skills to enhance resistance to substance use

(e.g., opposing peer pressure to use substances) (Paz Castro, et al., 2022).

4

Participation in life skills workshops provides an opportunity for drug addicts to

meet and communicate with others who have the same problem. The participants

can share their remedies and approaches to deal with drug abuse, avoid recurrence,

and handle cravings. They could provide multiparty support to improve the chance

of keeping away from the drug. Moreover, intra-network social supports are

against the sense of seclusion, isolation and foster interpersonal relationships

(Jahanbin, et al., 2017)

Nurses are well placed to serve a key role in teams seeking to help

individuals to avoid relapses. They often had critical knowledge about the

community resources and trends. Also, their ability to provide a wide range of

interventions ranging from supportive therapy to medical interventions often

proves to be an asset to patients (Guenzel & McChargue, 2022)

Substance use disorders are highly prevalent among youth and adult

populations. It is estimated that 10% of adolescents and between 20% and 30% of

adults (Centers for Disease Control CDC, 2021). The prevalence of substance use

disorders is 5.9% in Egypt, the population between 15-25 is the most exposed to

substance abuse and between 25-35 years is the most requested for treatment

(Addiction Treatment and Abuse Fund, 2022). Relapse rates after treatment have

been shown in other surveys to be as high as 40–75% in the 3 weeks to 6 months

following treatment (Moradinazar, et al., 2020).

The recovery (management and rehabilitation) processes from substance use

disorders are not inclusive enough and confine members to physical attendance for

the purpose of detoxification, neglecting the important factors such as life skills,

social, cultural, economic, environmental, and family factors. Since after

detoxification of the substances users return to their family and society, there can't

be expect a perfect quit without considering these factors carefully (Jepkorir,

2023).

Life skill educational program to enhance self-efficacy as a preventive

approach in which it focuses on the development of personal and social skills.

Previous studies revealed that there were few studies about the effects of life skills

training on relapse prevention among patients with substances use disorders

6

(Volkow, 2020). Therefore, the present study is an attempt to introduce a safe and

reasonable training program that help patients with substance use disorders to

enhance abstinence self-efficacy.

Aim of the study

The study aims: to evaluate the effect of life-skills training program on self-

efficacy among patients with substance use disorders.

The aim of this study will be achieved through the following objectives:

1- Assessing self-efficacy among patients with "substance use disorders".

2- Assessing risk for relapse among patients with "substance use disorders".

3- Developing life skills training program for self-efficacy among patients

with substance-use disorders based on identified their needs.

4- Implementing the developed life skills training program of relapse

prevention among patients with substance-use disorders.

5- Evaluating the effect of implementing life skills training program on self-

efficacy among patients with "substance-use disorders".

**Research Hypothesis** 

Life skills training program will have a positive effect on self-efficacy among patients with substance-use disorders.

### **Subjects & Methods**

#### Study design

A quasi-experimental research design on one group (pre-post) test will be used to conduct the current study.

## **Study setting**

The study will be conducted at Alabbasya Mental Health Hospital in Cairo. It is the oldest and biggest hospital for psychiatric illnesses in Egypt, affiliated to General Secretariat of Mental Health and Addiction Treatment of the Ministry of Health. It was established in 1883 A.D over an area of 68 acres. Its capacity is 1950 beds. The hospital structure is divided into such as, sections: Twenty-one old free sections, four illegal sections (forensic), two new buildings one of them for males that included addiction treatment and rehabilitation department in new building (2<sup>nd</sup> -3<sup>rd</sup> -4<sup>th</sup>) floor included detox ward about 30 bed, rehabilitation ward 60 bed, and dual ward, and another one for females. also, clinics such as, outpatient clinic - addiction clinic - children clinic - adolescent clinic - daycare

8

clinic - aging clinic - dental clinic - electroencephalogram clinic and electro

compulsive therapy clinic.

**Subjects** 

A purposive sample will be obtained from patients with "substances use

disorders" who meet inclusion criteria during their existence in the previously

mentioned setting.

Inclusion criteria:

- Age: from 20 years to 50 years.

- Had history of one episode of relapse

- Free from any physical disease such as diabetes, hypertension, viral

hepatitis etc.)

- Free from other Psychiatric disorders.

Sample size

Based on power analysis; Type I error ( $\alpha$ ) =0.05 with confidence level (1- $\alpha$ )

=0.95 and Type II error ( $\beta$ ) = 85%, by power test (1-  $\beta$ ) =0.15, sample size was

calculated according to the following equation that has been adopted from (Gupta, et al, 2016)

$$N=2(Z_{\alpha}+x_{[1-\beta]})^2\times SD^2/d^2$$

Where: n is the sample size,  $Z\alpha$  and Z (1- $\beta$ ) are constant values for convention values of  $\alpha$  and  $\beta$  values where  $Z\alpha$  =1.96 when  $\alpha$ =0.05 and Z (1- $\beta$ ) =1.036 when  $\beta$  =0.20, SD is the standard deviation obtained from previous study Moshki, et al., (2014) and d is the effect size.

$$N=2(1.96+1.03)^2 \times 7.7^2/5^2 = 42.4$$

Therefore, the minimal sample size was found to be =50 participants

Tools of data collection

# Tool I: Interview Questionnaire

It will be designed by the researcher and reviewed by supervisors. It will be written in the Arabic language for gathering data in relation to the following parts:

**Patients' characteristics**. such as age, marital status, residence, qualifications, starting and years of substance use.... etc.

Clinical data (addiction History). about substances as types of substance, onset, duration, route, etc.

## Tool II: Alcohol Abstinence Self-Efficacy Scale (AASE)

It was adapted by the researcher from DiClemente et al., (1994) to assess

10

personal confidence against taken substance. It consists of 40 items for assessing

self-efficacy. It includes 4 domain parts unranked: negative effect (1-5-9-13-17-21-

25-29-33-37), social/positive situations (2-6-10-14-18-22-26-30-34-38), physical

and other concern (3-7-11-15-19-23-27-31-35-39), and craving and urges(4-8-12-

16-20-24-28-32-36-38). Every domain includes 10 items.

Scoring system. Each statement was rated on 5 points as a Likert Skill Scale

ranged by statistical from (1) No Confidence, (2) Low Confidence, (3) Middle

Confidence, (4) High Confidence, and (5) Excellent Confidence. The total score

ranged from 40:200 ranged as, Low self-efficacy 40 < 120, Middle self-efficacy

121 < 160, and High self-efficacy 161 < 200.

Validity:

The one tool will be formulated and submitted to (5) experts in psychiatric and

mental health nursing or other specialty who will review the content of the tools

for their comprehensiveness, accuracy, clarity, and relevance.

Reliability:

Cronbach's Alpha will be used to determine the internal reliability of the tool.

**Preparatory Phase** 

This phase will be included reviewing of literature related to substance use

11

disorder, relapse prevention, this served study tools for data collection. During this

phase, the researcher also will be visited the selected place to be acquainted with

the staff and the study settings.

**Ethical considerations:** 

Research approval obtained from the faculty of Nursing- Ain Shams

University Ethical Committee before starting the study. The researcher explained

the aim and objectives of the study to patients with substance use disorder included

in the study before starting. Written approval obtained from patients with

substance use disorders before inclusion in the study. They guarantee that all the

gathered data will be used confidentially and will be used for research purposes

only. The researcher maintain anonymity and confidentiality of subjects' data

included in the study. Patients with substance use disorder will be informed that

they allow for withdrawal from study at any time.

Administrative design

Approval will be obtained through an issued letter from the dean of faculty of

nursing to directors of the previously mentioned setting. The researcher will be met

by the director to explain the purpose and methods of data collection and obtain

participants consent of share in the study after explain anything such as, related to

study and rights of withdrawal, free from harm. Data collected from the studied

sample will be revised, coded, and entered using a personal computer (PC).

Computerized data entry and statistical analysis will be conducted using the

statistical package for social sciences (SPSS).

Pilot study

The pilot study will be done on 10% (5 Patients) of the sample to examine

the clarity of tools and to estimate time needed to fill in the study tools. Based on

the results, modifications will be done (if necessary). Subjects included in the pilot

study will be excluded from the study if major modifications are required.

Field work

- The researcher will explain the aim of the study and the components of

the tools to the studied patients.

- The researcher will distribute a questionnaire to the studied patients to

assess their self-efficacy.

- The researcher will distribute a questionnaire to the patients studied to

assess the risk of relapse.

- The researcher trained patients in improving their life-skills.

**Life-skills Training Program** 

Life-Skills Training program will be developed by the researcher and

reviewed by supervisors for Enhance self-efficacy among patients with substance

use disorders. After reviewing the past and current related literature through

teaching the patients how to identify, plan and participate in relapse prevention.

The program will cover an overview of substance use disorders, relapse

prevention, self-efficacy, and many of life skills such as problems solving,

assertiveness, negotiation, refusal, time management, meditation, emotional

regulations, and non-violence communication skills.

Results

The results of the study will be presented in tables and figures that are easy to

understand and will be analyzed for inferring information and the proper

comments will be stated.

**Discussion** 

The results will be discussed in the light of available national and

international studies.

Conclusion

It will be derived from the finding of the study based on the research

hypothesis.

Recommendations

It will be derived from the discussion based on the findings of the study.

**Summary** 

It will include a brief description of the study process.

#### References

- Abdelmouttelb, A. A., Mahmoud, S., Elewa, M., & Abdelsalhen, F. A. (2022).

  Relation between substance use craving and self-efficacy in addict patients.

  Ekb.Eg. Retrieved March 17, 2023, from <a href="https://ejhc.journals.ekb.eg/article\_251533\_7a928fa6b43dc30ac7af5a49c960">https://ejhc.journals.ekb.eg/article\_251533\_7a928fa6b43dc30ac7af5a49c960</a>

  5e71.pdf
- Addiction Treatment and Abuse Fund (2022): prevalence of addiction and substance abuse in Egypt, <a href="https://mentalhealth.mohp.gov.eg/mental/web/sites/default/files/files/National%20survey%20report.pdf">https://mentalhealth.mohp.gov.eg/mental/web/sites/default/files/files/National%20survey%20report.pdf</a>
- Alanazi, A. M., Almutairi, S. F., Alsarami, A. A., Alanazi, F. J., Alqahtani, L. H., Alotaibi, T. F., ... & Ismaeil, T. T. (2022). Effects of Abstinence Self-Efficacy and Outcome Expectancies of Tobacco Smoking on the Desire to Quit Among Saudi Women: A Cross-Sectional Mediation Analysis. Tobacco Use

  Insights, vol 15, <a href="https://journals.sagepub.com/doi/full/10.1177/1179173X221075581">https://journals.sagepub.com/doi/full/10.1177/1179173X221075581</a>
- Bahramabadian, F., Mojtabaie, M., & Sabet, M. (2021). Comparison of the efficacy of acceptance and commitment-based therapy and schema therapy

- on self-efficacy and craving for change in addicts. Journal of psychological science. Vol, 20 issue 106 pp: 1849-1863
- CDC (2021) Wide-ranging online data for epidemiologic research (WONDER).

  Atlanta, GA, National Center for Health Statistics. Available at <a href="http://wonder.cdc.gov">http://wonder.cdc.gov</a>
- DiClemente, C.C., Carbonari, J.P., Montgomery, R.P.G. & Hughes, S.O. (1994). the Alcohol Abstinence Self-Efficacy Scale. Journal of Studies on Alcohol, 55, 141-148
- Ebrahem, S. M., Radwan, H. A., & El Amrosy, S. (2022). The effectiveness of life skills training on assertiveness, self-esteem, and aggressive behavior among patients with substance use disorders. International Egyptian Journal of Nursing Sciences and Research, 2(2), 413–431. https://doi.org/10.21608/ejnsr.2022.212482
- Guenzel, N., & McChargue, D. (2022). *Addiction Relapse Prevention*. StatPearls Publishing. <a href="https://doi.org/10.1186/s13011-021-00347-0">https://doi.org/10.1186/s13011-021-00347-0</a>
- Gupta, K., Attri, J., Singh, A., Kaur, H., & Kaur, G. (2016):

  Basic concepts for sample size calculation: Critical step for any clinical trials,

  Saudi J Anaesth, 10(3), 328-331.

- Jahanbin, I., Bazrafshan, M.-R., Akbari, K., Rahmati, M., & Ghadakpour, S. (2017). The effect of life skills training on social communication of clients referring to drug abuse clinics. Jundishapur Journal of Chronic Disease Care, In Press (In Press). https://doi.org/10.5812/jjcdc.13798
- Jepkorir, C. (2023). Effect of psychosocial interventions on management of adolescents risky behaviour in Therapeutic Communities in Uasin Gishu County, Kenya. The Catholic University of Eastern Africa.
- Miller, W. R., & Harris, R. J. (2000). A simple scale of Gorski's warning signs for relapse. Journal of Studies on Alcohol, 61, 759-765.
- Moradinazar, M., Farnia, V., Alikhani, M., Karyani, A. K., Rezaei, S., Rezaeian, S., Matin, B. K., & Najafi, F. (2020). Factors related to relapse in patients with substance-related disorders under methadone maintenance therapy:

  Decision tree analysis. Oman Medical Journal, 35(1), e89.

  <a href="https://doi.org/10.5001/omj.2020.07">https://doi.org/10.5001/omj.2020.07</a>
- Moshki, M., Hassanzade, T., & Taymoori, P. (2014). Effect of life skills training on drug abuse preventive behaviors among university students. *International Journal of Preventive Medicine*, *5*(5), 577–583.
- Niles, J. K., Gutierrez, D., Dukes, A. T., Mullen, P. R., & Goode, C. D. (2022). "Understanding the relationships between personal growth initiative, hope,

- and abstinence self-efficacy," *Journal of addictions & offender counseling*, 43(1), pp. 15–25. doi: 10.1002/jaoc.12099
- Paz Castro, R., Haug, S., Wenger, A., & Schaub, M. P. (2022). Longer-term efficacy of a digital life-skills training for substance use prevention.

  American Journal of Preventive Medicine, 63(6), 944–953.

  <a href="https://doi.org/10.1016/j.amepre.2022.06.017">https://doi.org/10.1016/j.amepre.2022.06.017</a>
- Sapkota, S., Khadka, A., & Akela, G. (2019). Contributing factors to relapse of drug addiction among clients attending rehabilitation centres of Dharan, Nepal. *Journal of Chitwan Medical College*, 6(3), 20–25. <a href="https://doi.org/10.3126/jcmc.v6i3.16695">https://doi.org/10.3126/jcmc.v6i3.16695</a>
- Unicef.org. Retrieved March 12, 2023, from, <a href="https://www.unicef.org/azerbaijan/media/1541/file/basic%20life%20skills.pd">https://www.unicef.org/azerbaijan/media/1541/file/basic%20life%20skills.pd</a> <a href="mailto:file/basic%20life%20skills.pd">f</a>
- Unodc.org. (2023). Module 7 Life Skills. Retrieved March 12, 2023, from <a href="https://www.unodc.org/pdf/youthnet/action/message/escap\_peers\_07.pdf">https://www.unodc.org/pdf/youthnet/action/message/escap\_peers\_07.pdf</a>
- Volkow, D. N., (2020). Drugs, Brain, Behavior: The Science of Addiction.

  National Institute for Drug Abuse. Science of Addiction, 7(3), 1–32.

  <a href="https://www.drugabuse.gov/publications/drugs-brains-behavior-science-addiction/drugs-brain">https://www.drugabuse.gov/publications/drugs-brains-behavior-science-addiction/drugs-brain</a>

WHO (2023). Life skills education planning for research division of mental health and prevention of substance abuse. Retrieved March 12, 2023, from <a href="https://apps.who.int/iris/bitstream/handle/10665/338491/MNH-PSF-96.2.Rev.1-eng.pdf">https://apps.who.int/iris/bitstream/handle/10665/338491/MNH-PSF-96.2.Rev.1-eng.pdf</a>